CLINICAL TRIAL: NCT04171141
Title: A PHASE 1 DOSE ESCALATION AND EXPANSION STUDY EVALUATING THE SAFETY, TOLERABILITY, PHARMACOKINETICS, PHARMACODYNAMICS AND ANTI TUMOR ACTIVITY OF PF-07062119 IN PATIENTS WITH ADVANCED GASTROINTESTINAL TUMORS
Brief Title: Study to Test the Safety and Tolerability of PF-07062119 in Patients With Selected Advanced or Metastatic Gastrointestinal Tumors.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated due to strategic considerations and not due to safety.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C3861001; GUCY2C (Other: Alias Study Number)
Record Dates: First submitted 2019-11-08; First posted 2019-11-20 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Gastrointestinal Tumors; Colorectal Adenocarcinomas; Gastric Adenocarcinomas; Esophageal Adenocarcinomas
Keywords: Gastric cancer; Esophageal cancer; Colorectal cancer; Advanced esophageal cancer; Metastatic esophageal cancer; Advanced colorectal cancer; Metastatic gastric cancer; Advanced gastric cancer; Metastatic colorectal cancer; GUCY2c; Anti-PD1; Anti-VEGF; Measurable disease; PF-07062119; PF-06801591; Bevacizumab
MeSH Terms: conditions — Digestive System Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Colorectal Neoplasms | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Dose Escalation (Experimental): Single Agent Dose Escalation
  Interventions: Drug: PF-07062119
- Dose Finding Anti-PD-1 Combination (Experimental): Part 1B PF-07062119 plus anti-PD-1
  Interventions: Drug: PF-07062119; Drug: Anti-PD1
- Dose Finding anti-VEGF Combination (Experimental): Part 1B PF-07062119 plus anti-VEGF
  Interventions: Drug: PF-07062119; Drug: Anti-VEGF
- Dose Expansion Arm A (Experimental): PF-07062119 as a Single Agent in CRC
  Interventions: Drug: PF-07062119
- Dose Expansion Arm B (Experimental): PF-07062119 in Combination with anti-PD-1 in CRC
  Interventions: Drug: PF-07062119
- Dose Expansion Arm C (Experimental): PF-07062119 in Combination with anti-VEGF in CRC
  Interventions: Drug: PF-07062119; Drug: Anti-PD1; Drug: Anti-VEGF
- Dose Expansion Arm D (Experimental): PF-07062119 in Combination with either anti-PD-1 or anti-VEGF in various Tumor Types
  Interventions: Drug: PF-07062119; Drug: Anti-PD1; Drug: Anti-VEGF

INTERVENTIONS:
Drug: PF-07062119 — PF-07062119
Drug: Anti-PD1 — Anti-PD1 PF-06801591
  Arms: Dose Expansion Arm C; Dose Expansion Arm D; Dose Finding Anti-PD-1 Combination
Drug: Anti-VEGF — Anti-VEGF IV (bevacizumab)
  Arms: Dose Expansion Arm C; Dose Expansion Arm D; Dose Finding anti-VEGF Combination

SUMMARY:
A phase 1, open-label, dose escalation and expansion study of PF-07062119 in patients with selected advanced or metastatic gastrointestinal tumors

DETAILED DESCRIPTION:
This is a Phase 1, open-label, multi-center, non-randomized, multiple dose, safety, tolerability, pharmacokinetic, and pharmacodynamic study of PF-07062119 administered as a single agent in sequential dose levels and then in combination with anti-programmed cell death -1 protein (anti-PD-1) and in combination with an anti-vascular endothelial growth factor (anti-VEGF). In Part 1A, successive cohorts of patients will receive escalating doses of PF-007062119 and then in dose finding (Part 1B) with PF-07062119 in combination with anti-PD-1 and in combination with anti-VEGF. This study contains 2 parts, dose escalation with single agent (Part 1A) and then dose finding with PF-007062119 in combination with ant-PD-1 and in combination with anti-VEGF (Part 1B) followed by dose expansion arms as a single agent and PF-07062119 in combination with anti-PD 1 and in combination with anti-VEGF (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* For Part 1 and Part 2, diagnosis of advanced/metastatic colorectal, gastric or esophageal adenocarcinoma that is resistant to standard therapy or for which no local regulatory approved standard therapy is available that would confer significant benefit.
* For Part 2, diagnosis of colorectal adenocarcinoma that is resistant to standard therapy or for which no standard therapy is available
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1
* Measurable disease or non-measurable disease and refractory to or intolerant of existing therapies (Part 1)
* Measurable disease as defined by RECIST 1.1 is required (Part 2)

Exclusion Criteria:

* Known active uncontrolled or symptomatic Central Nervous System (CNS) metastases
* Other active malignancy within 3 years prior to randomization, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ
* Major surgery or radiation within 3 weeks prior to study entry
* Last anti-cancer treatment within 4 weeks prior to study entry
* Active or history of clinically significant autoimmune disease that required systemic immunosuppressive medication
* Active or history of clinically significant gastrointestinal disease
* Participation in other studies involving investigational drug(s) within 2 weeks prior to study entry
* Pregnant or breastfeeding female patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- United States (15):
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - City of Hope IDS Pharmacy, Duarte, California
  - UCLA Department of Medicine: Hematology-Oncology, Los Angeles, California
  - UCLA Hematology Oncology - Santa Monica, Santa Monica, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Inpatient Pavilion (AIP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Outpatient Pavilion (AOP), Aurora, Colorado
  - START Midwest, Grand Rapids, Michigan
  - Memorial Sloan Kettering Cancer Center Rockefeller Outpatient Pavillion, New York, New York
  - Evelyn H. Lauder Breast and Imaging Center, New York, New York
  - Memorial Sloan Kettering Cancer Center - Main Campus, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Christus Santa Rosa Hospital, San Antonio, Texas
  - NEXT Oncology, San Antonio, Texas
- Australia (2):
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Cancer Center Hospital, Chuo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3861001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dose Expansion Phase (Part 2) of the study was not conducted due to the study termination. Study termination was due to a strategic decision but not any safety concerns or requests from any regulatory authorities.
Groups:
- Part 1A PF-07062119 45 µg: Participants received PF-07062119 45 µg via subcutaneous (SC) injection as monotherapy every 2 weeks (Q2W) at every cycle (1 cycle=28 days) without a priming dose.
- Part 1A PF-07062119 135 µg: Participants received PF-07062119 135 µg via SC injection as monotherapy Q2W at every cycle (1 cycle=28 days) without a priming dose.
- Part 1A PF-07062119 400 µg: Participants received PF-07062119 400 µg via SC injection as monotherapy Q2W at every cycle (1 cycle=28 days) without a priming dose.
- Part 1A PF-07062119 800 µg: Participants received PF-07062119 800 µg via SC injection as monotherapy Q2W at every cycle (1 cycle=28 days) without a priming dose.
- Part 1A PF-07062119 1600 µg: Participants received PF-07062119 1600 µg via SC injection as monotherapy without a priming dose Q2W at every cycle (1 cycle=28 days).
- Part 1A PF-07062119 400 µg/800 µg: Participants received a priming dose of PF-07062119 400 µg on Cycle 1 Day 1 via SC injection, followed by a full dose of 800 µg Q2W since Cycle 1 Day 15.
- Part 1A PF-07062119 400 µg/1200 µg: Participants received a priming dose of PF-07062119 400 µg on Cycle 1 Day 1 via SC injection, followed by a full dose of 1200 µg Q2W since Cycle 1 Day 15.
- Part 1A PF-07062119 400 µg/1600 µg: Participants received a priming dose of PF-07062119 400 µg on Cycle 1 Day 1 via SC injection, followed by a full dose of 1600 µg Q2W since Cycle 1 Day 15.
- Part 1A PF-07062119 400 µg/2100 µg: Participants received a priming dose of PF-07062119 400 µg on Cycle 1 Day 1 via SC injection, followed by a full dose of 2100 µg Q2W since Cycle 1 Day 15.
- Part 1A PF-07062119 400 µg/2800 µg: Participants received a priming dose of PF-07062119 400 µg on Cycle 1 Day 1 via SC injection, followed by a full dose of 2800 µg Q2W since Cycle 1 Day 15.
- Part 1A PF-07062119 400 µg/3700 µg: Participants received a priming dose of PF-07062119 400 µg on Cycle 1 Day 1 via SC injection, followed by a full dose of 3700 µg Q2W since Cycle 1 Day 15.
- Part 1B PF-07062119 400 µg Q2W + PF-06801591 300 mg Q4W: Participants received PF-07062119 400 µg Q2W + PF-06801591 300 mg (50 mg/mL) every 4 weeks (Q4W) via SC injection.
- Part 1B PF-07062119 800 µg Q2W + PF-06801591 300 mg Q4W-Priming: Participants received PF-07062119 800 µg Q2W + PF-06801591 300 mg (50 mg/mL) Q4W via SC injection.
- Part 1B PF-07062119 1200 µg Q2W + PF-06801591 300 mg Q4W-Priming: Participants received PF-07062119 1200 µg Q2W + PF-06801591 300 mg (50 mg/mL) Q4W via SC injection.
- Part 1B PF-07062119 800 µg Q2W + Bevacizumab 5 mg/kg Q2W: Participants received PF-07062119 800 µg Q2W via SC injection + bevacizumab-Pfizer via intravenous (IV) infusion Q2W based on 5 mg/kg of body weight.
- Part 1B PF-07062119 1200 µg Q2W + Bevacizumab 5 mg/kg Q2W-Priming: Participants received PF-07062119 1200 µg Q2W via SC injection + bevacizumab-Pfizer via IV infusion Q2W based on 5 mg/kg of body weight.
Period: Overall Study
Arm/Group | Part 1A PF-07062119 45 µg | Part 1A PF-07062119 135 µg | Part 1A PF-07062119 400 µg | Part 1A PF-07062119 800 µg | Part 1A PF-07062119 1600 µg | Part 1A PF-07062119 400 µg/800 µg | Part 1A PF-07062119 400 µg/1200 µg | Part 1A PF-07062119 400 µg/1600 µg | Part 1A PF-07062119 400 µg/2100 µg | Part 1A PF-07062119 400 µg/2800 µg | Part 1A PF-07062119 400 µg/3700 µg | Part 1B PF-07062119 400 µg Q2W + PF-06801591 300 mg Q4W | Part 1B PF-07062119 800 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 800 µg Q2W + Bevacizumab 5 mg/kg Q2W | Part 1B PF-07062119 1200 µg Q2W + Bevacizumab 5 mg/kg Q2W-Priming
Started | 2 | 3 | 6 | 9 | 2 | 10 | 6 | 6 | 8 | 4 | 4 | 3 | 4 | 4 | 5 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 3 | 6 | 9 | 2 | 10 | 6 | 6 | 8 | 4 | 4 | 3 | 4 | 4 | 5 | 3
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Progressive disease | 2 | 3 | 4 | 7 | 1 | 8 | 4 | 6 | 7 | 3 | 4 | 3 | 4 | 2 | 4 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Global deterioration of health status | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who received at least 1 dose of randomized study medication and had a baseline and at least 1 post-baseline measurement (after taking randomization study medication).
Groups:
- Part 1A PF-07062119 1600 µg: Participants received PF-07062119 1600 µg via subcutaneous (SC) injection as monotherapy without a priming dose Q2W at every cycle (1 cycle=28 days).
- Total: Total of all reporting groups
Arm/Group | Part 1A PF-07062119 45 µg | Part 1A PF-07062119 135 µg | Part 1A PF-07062119 400 µg | Part 1A PF-07062119 800 µg | Part 1A PF-07062119 1600 µg | Part 1A PF-07062119 400 µg/800 µg | Part 1A PF-07062119 400 µg/1200 µg | Part 1A PF-07062119 400 µg/1600 µg | Part 1A PF-07062119 400 µg/2100 µg | Part 1A PF-07062119 400 µg/2800 µg | PART 1A PF-07062119 400 µg/3700 µg | Part 1B PF-07062119 400 µg Q2W + PF-06801591 300 mg Q4W | Part 1B PF-07062119 800 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 800 µg Q2W + Bevacizumab 5 mg/kg Q2W | Part 1B PF-07062119 1200 µg Q2W + Bevacizumab 5 mg/kg Q2W-Priming | Total
Number analyzed (Participants) | 2 | 3 | 6 | 9 | 2 | 10 | 6 | 6 | 8 | 4 | 4 | 3 | 4 | 4 | 5 | 3 | 79
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64 (16.97) | 60.7 (6.03) | 60.8 (10.38) | 56.9 (10.97) | 41.0 (12.73) | 55.9 (15.49) | 63.3 (15.36) | 55.2 (13.11) | 55.5 (8.62) | 65.0 (11.34) | 62.3 (8.54) | 50.3 (9.61) | 53.3 (14.24) | 54.3 (18.80) | 52.2 (11.69) | 53.3 (9.61) | 56.9 (12.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 4 | 4 | 0 | 4 | 3 | 1 | 3 | 1 | 1 | 0 | 2 | 1 | 1 | 2 | 30
  Male | 1 | 1 | 2 | 5 | 2 | 6 | 3 | 5 | 5 | 3 | 3 | 3 | 2 | 3 | 4 | 1 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 12
  Not Hispanic or Latino | 1 | 1 | 4 | 8 | 1 | 8 | 6 | 5 | 6 | 3 | 4 | 1 | 4 | 3 | 5 | 2 | 62
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 4 | 0 | 3 | 2 | 1 | 4 | 2 | 2 | 0 | 2 | 1 | 1 | 0 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3
  White | 0 | 2 | 4 | 5 | 2 | 6 | 2 | 4 | 4 | 2 | 2 | 1 | 2 | 3 | 4 | 3 | 46
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) Assessed Through Cycle 1
Description: Hematological DLTs:
  * Grade 3 neutropenia lasting >5 days
  * Febrile neutropenia defined as an ANC <1.0 x 10 ̂9/L with a single temperature of >38.3°C, or a sustained temperature of ≥38°C, for more than 1 hour
  * Grade ≥3 Neutropenia with infection
  * Grade 3 Thrombocytopenia with Grade ≥2 (clinically significant) bleeding
  * any Grade 4 Thrombocytopenia
  * Anemia or Thrombocytopenia requiring transfusion
  Non Hematological DLTs:
  * Grade ≥3 fatigue lasting ≥7 days
  * for participants with liver, bone, or lung metastasis, an AST or ALT increase >8 x ULN or ALP >10 x ULN;
  * confirmed DILI meeting Hy's law criteria
  * Grade 3 Vomiting or Diarrhea lasting ≥3 days despite adequate treatment/other supportive care
  * Grade 4 Vomiting or Diarrhea
  * Grade ≥3 CRS regardless of duration
  * Grade ≥3 QTcF prolongation irrespective of duration
  * any death not clearly due to underlying disease or extraneous causes Clinically important/persistent toxicities were DLTs reviewed by investigators and sponsor.
Time Frame: 28 Days
Population: Analysis population included all enrolled participants who had at least 1 dose of study intervention and either experienced DLT or did not have major treatment deviations during the DLT observation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A PF-07062119 45 µg | Part 1A PF-07062119 135 µg | Part 1A PF-07062119 400 µg | Part 1A PF-07062119 800 µg | Part 1A PF-07062119 1600 µg | Part 1A PF-07062119 400 µg/800 µg | Part 1A PF-07062119 400 µg/1200 µg | Part 1A PF-07062119 400 µg/1600 µg | Part 1A PF-07062119 400 µg/2100 µg | Part 1A PF-07062119 400 µg/2800 µg | Part 1A PF-07062119 400 µg/3700 µg | Part 1B PF-07062119 400 µg Q2W + PF-06801591 300 mg Q4W | Part 1B PF-07062119 800 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 800 µg Q2W + Bevacizumab 5 mg/kg Q2W | Part 1B PF-07062119 1200 µg Q2W + Bevacizumab 5 mg/kg Q2W-Priming
Number analyzed (Participants) | 2 | 3 | 5 | 9 | 2 | 6 | 3 | 4 | 7 | 3 | 2 | 3 | 4 | 2 | 5 | 3
Participants | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With All-Causality Treatment-Emergent Adverse Events (TEAEs),Treatment-Emergent Serious Adverse Events (TESAEs), Maximum Grade 3 or 4 and 5 TEAEs
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was defined as any untoward medical occurrence that, at any dose: resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent disability/incapacity; was a congenital anomaly/birth defect, etc. Treatment-emergent events were with onset date occurring during the on-treatment period. AEs were documented and recorded at each visit using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.
Time Frame: 4 Years
Population: Analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A PF-07062119 45 µg | Part 1A PF-07062119 135 µg | Part 1A PF-07062119 400 µg | Part 1A PF-07062119 800 µg | Part 1A PF-07062119 1600 µg | Part 1A PF-07062119 400 µg/800 µg | Part 1A PF-07062119 400 µg/1200 µg | Part 1A PF-07062119 400 µg/1600 µg | Part 1A PF-07062119 400 µg/2100 µg | Part 1A PF-07062119 400 µg/2800 µg | PART 1A PF-07062119 400 µg/3700 µg | Part 1B PF-07062119 400 µg Q2W + PF-06801591 300 mg Q4W | Part 1B PF-07062119 800 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 800 µg Q2W + Bevacizumab 5 mg/kg Q2W | Part 1B PF-07062119 1200 µg Q2W + Bevacizumab 5 mg/kg Q2W-Priming
Number analyzed (Participants) | 2 | 3 | 6 | 9 | 2 | 10 | 6 | 6 | 8 | 4 | 4 | 3 | 4 | 4 | 5 | 3
Participants
  Number of Participants With All-Causality TEAEs | 2 | 3 | 6 | 9 | 2 | 10 | 6 | 6 | 8 | 4 | 4 | 3 | 4 | 4 | 5 | 3
  Number of Participants With All-Causality TESAEs | 0 | 1 | 2 | 3 | 1 | 4 | 4 | 2 | 4 | 1 | 2 | 0 | 0 | 3 | 2 | 1
  Number of Participants With Maximum Grade 3 or 4 TEAEs | 0 | 1 | 3 | 4 | 2 | 6 | 2 | 3 | 6 | 3 | 3 | 1 | 1 | 4 | 2 | 1
  Number of Participants With Maximum Grade 5 TEAEs | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Treatment-Related TEAEs, TESAEs, Maximum Grade 3 or 4 and 5 TEAEs
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was defined as any untoward medical occurrence that, at any dose: resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent disability/incapacity; was a congenital anomaly/birth defect, etc. Treatment-emergent events were with onset date occurring during the on-treatment period. Relatedness to study treatment was determined by the investigator. AEs were documented and recorded at each visit using the NCI CTCAE version 5.0. Severe AEs were classified as Grade 3; life-threatening consequences and urgent intervention indicated were classified as Grade 4; deaths related to AEs were classified as Grade 5.
Time Frame: 4 Years
Population: Analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A PF-07062119 45 µg | Part 1A PF-07062119 135 µg | Part 1A PF-07062119 400 µg | Part 1A PF-07062119 800 µg | Part 1A PF-07062119 1600 µg | Part 1A PF-07062119 400 µg/800 µg | Part 1A PF-07062119 400 µg/1200 µg | Part 1A PF-07062119 400 µg/1600 µg | Part 1A PF-07062119 400 µg/2100 µg | Part 1A PF-07062119 400 µg/2800 µg | Part 1A PF-07062119 400 µg/3700 µg | Part 1B PF-07062119 400 µg Q2W + PF-06801591 300 mg Q4W | Part 1B PF-07062119 800 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 800 µg Q2W + Bevacizumab 5 mg/kg Q2W | Part 1B PF-07062119 1200 µg Q2W + Bevacizumab 5 mg/kg Q2W-Priming
Number analyzed (Participants) | 2 | 3 | 6 | 9 | 2 | 10 | 6 | 6 | 8 | 4 | 4 | 3 | 4 | 4 | 5 | 3
Participants
  Number of Participants With Treatment-Related TEAEs | 2 | 3 | 6 | 9 | 2 | 10 | 6 | 6 | 8 | 4 | 4 | 3 | 4 | 4 | 5 | 3
  Number of Participants With Treatment-Related TESAEs | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 0 | 3 | 1 | 1 | 0 | 0 | 1 | 1 | 1
  Number of Participants With Treatment-Related Maximum Grade 3 or 4 TEAEs | 0 | 0 | 1 | 3 | 2 | 5 | 0 | 3 | 4 | 1 | 2 | 0 | 1 | 2 | 2 | 1
  Number of Participants With Treatment-Related Maximum Grade 5 TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With CTCAE Grade 3 or 4 Hematology Laboratory Abnormalities
Description: The investigator reviewed the laboratory report, documented this review, and recorded any clinically relevant changes occurring during the study in the AE section of the CRF. Clinically significant abnormal laboratory findings were those which were not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. CTCAE version 5.0 was applied.
Time Frame: 4 Years
Population: Analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A PF-07062119 45 µg | Part 1A PF-07062119 135 µg | Part 1A PF-07062119 400 µg | Part 1A PF-07062119 800 µg | Part 1A PF-07062119 1600 µg | Part 1A PF-07062119 400 µg/800 µg | Part 1A PF-07062119 400 µg/1200 µg | Part 1A PF-07062119 400 µg/1600 µg | Part 1A PF-07062119 400 µg/2100 µg | Part 1A PF-07062119 400 µg/2800 µg | Part 1A PF-07062119 400 µg/3700 µg | Part 1B PF-07062119 400 µg Q2W + PF-06801591 300 mg Q4W | Part 1B PF-07062119 800 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 800 µg Q2W + Bevacizumab 5 mg/kg Q2W | Part 1B PF-07062119 1200 µg Q2W + Bevacizumab 5 mg/kg Q2W-Priming
Number analyzed (Participants) | 2 | 3 | 6 | 9 | 2 | 10 | 6 | 6 | 8 | 4 | 4 | 3 | 4 | 4 | 5 | 3
Participants
  Grade 3 Lymphocyte count decreased | 0 | 1 | 2 | 1 | 1 | 3 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 0
  Grade 4 Lymphocyte count decreased | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Anemia | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 3 Hemoglobin increased | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Grade 3 White blood cell decreased | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 4 Platelet count decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With CTCAE Grade 3 or 4 Chemistry Laboratory Abnormalities
Description: The investigator reviewed the laboratory report, documented this review, and recorded any clinically relevant changes occurring during the study in the AE section of the case report form (CRF). Clinically significant abnormal laboratory findings were those which were not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. CTCAE version 5.0 was applied.
Time Frame: 4 Years
Population: Analysis population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A PF-07062119 45 µg | Part 1A PF-07062119 135 µg | Part 1A PF-07062119 400 µg | Part 1A PF-07062119 800 µg | Part 1A PF-07062119 1600 µg | Part 1A PF-07062119 400 µg/800 µg | Part 1A PF-07062119 400 µg/1200 µg | Part 1A PF-07062119 400 µg/1600 µg | Part 1A PF-07062119 400 µg/2100 µg | Part 1A PF-07062119 400 µg/2800 µg | Part 1A PF-07062119 400 µg/3700 µg | Part 1B PF-07062119 400 µg Q2W + PF-06801591 300 mg Q4W | Part 1B PF-07062119 800 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 800 µg Q2W + Bevacizumab 5 mg/kg Q2W | Part 1B PF-07062119 1200 µg Q2W + Bevacizumab 5 mg/kg Q2W-Priming
Number analyzed (Participants) | 2 | 3 | 6 | 9 | 2 | 10 | 6 | 6 | 8 | 4 | 4 | 3 | 4 | 4 | 5 | 3
Participants
  Grade 3 Alanine aminotransferase increased | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Alkaline phosphatase increased | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Aspartate aminotransferase increased | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 Aspartate aminotransferase increased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Blood bilirubin increased | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Grade 4 Blood bilirubin increased | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Creatinine increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 3 Hypermagnesemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Hypokalemia | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Grade 4 Hypomagnesemia | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Hyponatremia | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Lipase increased | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0
  Grade 4 Lipase increased | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0
  Grade 3 Serum amylase increased | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Grade 4 Serum amylase increased | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Cycle 1 and Cycle 4 PF-07062119 PK Parameters: Maximum Concentration (Cmax) - Priming Cohorts
Description: Cmax was observed directly from data.
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 4 Day 1
Population: Number of participants analyzed included all enrolled participants treated with at least 1 PK parameter of interest. Number analyzed refers to number of participants who had PK parameter results with no dose interruption/reduction before or on this visit.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1A PF-07062119 400 µg/800 µg | Part 1A PF-07062119 400 µg/1200 µg | Part 1A PF-07062119 400 µg/1600 µg | Part 1A PF-07062119 400 µg/2100 µg | Part 1A PF-07062119 400 µg/2800 µg | PART 1A PF-07062119 400 µg/3700 µg | Part 1B PF-07062119 800 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + Bevacizumab 5 mg/kg Q2W-Priming
Number analyzed (Participants) | 10 | 6 | 6 | 8 | 4 | 4 | 4 | 4 | 3
ng/mL
  Cycle 1 Day 1 | 27.75 (52) | 23.66 (33) | 30.98 (31) | 37.79 (53) | 36.04 (16) | 38.10 (16) | 29.32 (44) | 37.59 (31) | 37.37 (13)
  Cycle 1 Day 15: number analyzed (Participants) | 9 | 6 | 6 | 8 | 4 | 4 | 4 | 3 | 3
  Cycle 1 Day 15 | 67.03 (35) | 67.34 (53) | 142.1 (54) | 224.2 (59) | 333.9 (30) | 427.5 (6) | 76.74 (31) | 92.64 (60) | 143.2 (15)
  Cycle 4 Day 1: number analyzed (Participants) | 1 | 1 | 0 | 4 | 2 | 1 | 3 | 0 | 2
  Cycle 4 Day 1 | 145 (NA) — One participant with evaluable Cmax result at this visit, so the individual value is presented. | 190 (NA) — One participant with evaluable Cmax result at this visit, so the individual value is presented. |  | 598.1 (16) | 744.5 (NA) — Two participants with evaluable Cmax results at this visit (738 and 751 ng/mL), so the geometric %CV was NA. | 987 (NA) — One participant with evaluable Cmax result at this visit, so the individual value is presented. | 26.45 (13966) |  | 326.26 (NA) — Two participants with evaluable Cmax results at this visit (299 and 356 ng/mL), so the geometric %CV was NA.

7. Secondary Outcome: Cycle 1 and Cycle 4 PF-07062119 PK Parameters: Cmax - Non-Priming Cohorts
Description: Cmax was observed directly from data.
Time Frame: Cycle 1 Day 1 and Cycle 4 Day 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1A PF-07062119 45 µg | Part 1A PF-07062119 135 µg | Part 1A PF-07062119 400 µg | Part 1A PF-07062119 800 µg | Part 1A PF-07062119 1600 µg | Part 1B PF-07062119 400 µg Q2W + PF-06801591 300 mg Q4W | Part 1B PF-07062119 800 µg Q2W + Bevacizumab 5 mg/kg Q2W
Number analyzed (Participants) | 2 | 3 | 6 | 9 | 2 | 3 | 5
ng/mL
  Cycle 1 Day 1 | 2.96 (NA) — Two participants with evaluable Cmax results at this visit (2.93 and 3.00 ng/mL), so the geometric %CV was NA. | 9.032 (10) | 43.67 (40) | 66.75 (39) | 132.2 (NA) — Two participants with evaluable Cmax results at this visit (115 and 152 ng/mL), so the geometric %CV was NA. | 23.35 (16) | 55.96 (29)
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1 | 1
  Cycle 4 Day 1 |  |  | 110 (NA) — One participant with evaluable Cmax result at this visit, so the individual value is presented. | 164.92 (NA) — Two participants with evaluable Cmax results at this visit (136 and 200 ng/mL), so the geometric %CV was NA. |  | 62.9 (NA) — One participant with evaluable Cmax result at this visit, so the individual value is presented. | 193 (NA) — One participant with evaluable Cmax result at this visit, so the individual value is presented.

8. Secondary Outcome: Cycle 1 and Cycle 4 PF-07062119 PK Parameters: Time to Achieve Cmax (Tmax) - Priming Cohorts
Description: Tmax was time at which Cmax occurred which was observed directly from data as time of first occurrence.
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 4 Day 1
Population: as for outcome 6
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 1A PF-07062119 400 µg/800 µg | Part 1A PF-07062119 400 µg/1200 µg | Part 1A PF-07062119 400 µg/1600 µg | Part 1A PF-07062119 400 µg/2100 µg | Part 1A PF-07062119 400 µg/2800 µg | PART 1A PF-07062119 400 µg/3700 µg | Part 1B PF-07062119 800 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + Bevacizumab 5 mg/kg Q2W-Priming
Number analyzed (Participants) | 10 | 6 | 6 | 8 | 4 | 4 | 4 | 4 | 3
Hour
  Cycle 1 Day 1 | 167 [152 to 360] | 222 [141 to 335] | 178 [144 to 332] | 165 [143 to 386] | 167 [164 to 187] | 167 [144 to 192] | 167 [23.4 to 330] | 167 [164 to 190] | 166 [164 to 190]
  Cycle 1 Day 15: number analyzed (Participants) | 9 | 6 | 6 | 8 | 4 | 4 | 4 | 3 | 3
  Cycle 1 Day 15 | 162 [94.0 to 187] | 129 [21.7 to 214] | 152 [88.1 to 192] | 151 [89.6 to 192] | 128 [8.88 to 168] | 132 [72.4 to 171] | 111 [94.7 to 167] | 167 [23.9 to 170] | 73.2 [46.2 to 163]
  Cycle 4 Day 1: number analyzed (Participants) | 1 | 1 | 0 | 4 | 2 | 1 | 3 | 0 | 2
  Cycle 4 Day 1 | 19.0 [19.0 to 19.0] | 21.8 [21.8 to 21.8] |  | 83.5 [25.3 to 209] | 131 [118 to 144] | 26.5 [26.5 to 26.5] | 94.5 [18.2 to 140] |  | 104.2 [67.4 to 141]

9. Secondary Outcome: Cycle 1 and Cycle 4 PF-07062119 PK Parameters: Tmax - Non-Priming Cohorts
Description: Tmax was time at which Cmax occurred which was observed directly from data as time of first occurrence.
Time Frame: Cycle 1 Day 1 and Cycle 4 Day 1
Population: as for outcome 6
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 1A PF-07062119 45 µg | Part 1A PF-07062119 135 µg | Part 1A PF-07062119 400 µg | Part 1A PF-07062119 800 µg | Part 1A PF-07062119 1600 µg | Part 1B PF-07062119 400 µg Q2W + PF-06801591 300 mg Q4W | Part 1B PF-07062119 800 µg Q2W + Bevacizumab 5 mg/kg Q2W
Number analyzed (Participants) | 2 | 3 | 6 | 9 | 2 | 3 | 5
Hour
  Cycle 1 Day 1 | 173.11 [8.22 to 338] | 186 [94.7 to 191] | 93.3 [90.7 to 387] | 96.8 [26.0 to 192] | 35.85 [23.7 to 48.0] | 170 [96.5 to 187] | 94.0 [46.2 to 383]
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 0 | 1 | 1
  Cycle 4 Day 1 |  |  | 95.4 [95.4 to 95.4] | 95.5 [24.0 to 167] |  | 96.2 [96.2 to 96.2] | 23.4 [23.4 to 23.4]

10. Secondary Outcome: Cycle 1 and Cycle 4 PF-07062119 PK Parameters: Area Under the Serum Concentration-Time Profile From Time 0 to Time Tau, the Dosing Interval (AUCtau) - Priming Cohorts
Description: AUCtau was area under the serum concentration-time profile from time 0 to time tau, the dosing interval, determined using linear/Log trapezoidal method.
Time Frame: Cycle 1 Day 1 and Cycle 4 Day 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hour/mL
Arm/Group | Part 1A PF-07062119 400 µg/800 µg | Part 1A PF-07062119 400 µg/1200 µg | Part 1A PF-07062119 400 µg/1600 µg | Part 1A PF-07062119 400 µg/2100 µg | Part 1A PF-07062119 400 µg/2800 µg | PART 1A PF-07062119 400 µg/3700 µg | Part 1B PF-07062119 800 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + Bevacizumab 5 mg/kg Q2W-Priming
Number analyzed (Participants) | 10 | 6 | 6 | 8 | 4 | 4 | 4 | 4 | 3
ng•hour/mL
  Cycle 1 Day 1 | 6527 (38) | 5612 (43) | 7864 (42) | 9712 (52) | 9169 (14) | 10030 (19) | 8387 (37) | 9233 (37) | 8887 (13)
  Cycle 4 Day 1: number analyzed (Participants) | 1 | 1 | 0 | 4 | 2 | 1 | 3 | 0 | 2
  Cycle 4 Day 1 | 42300 (NA) — There was 1 evaluable AUCtau measurement at this visit. | 60200 (NA) — There was 1 evaluable AUCtau measurement at this visit. |  | 168000 (NA) — There was 1 evaluable AUCtau measurement at this visit. | 210000 (NA) — There was 1 evaluable AUCtau measurement at this visit. | 304000 (NA) — There was 1 evaluable AUCtau measurement at this visit. | 32500 (NA) — There was 1 evaluable AUCtau measurement at this visit. |  | 89600 (NA) — There was 1 evaluable AUCtau measurement at this visit.

11. Secondary Outcome: Cycle 1 and Cycle 4 PF-07062119 PK Parameters: AUCtau - Non-Priming Cohorts
Description: as for outcome 10
Time Frame: Cycle 1 Day 1 and Cycle 4 Day 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hour/mL
Arm/Group | Part 1A PF-07062119 45 µg | Part 1A PF-07062119 135 µg | Part 1A PF-07062119 400 µg | Part 1A PF-07062119 800 µg | Part 1A PF-07062119 1600 µg | Part 1B PF-07062119 400 µg Q2W + PF-06801591 300 mg Q4W | Part 1B PF-07062119 800 µg Q2W + Bevacizumab 5 mg/kg Q2W
Number analyzed (Participants) | 2 | 3 | 6 | 9 | 2 | 3 | 5
ng•hour/mL
  Cycle 1 Day 1 | 802.577 (NA) — Two participants with evaluable AUCtau results at this visit (765 and 842 ng•hour/mL), so the geometric %CV was NA. | 2618 (8) | 12060 (43) | 19120 (35) | NA (NA) — No participant had evaluable AUCtau result at this visit. | 6346.2 (NA) — Two participants with evaluable AUCtau results at this visit (5170 and 7790 ng•hour/mL), so the geometric %CV was NA. | 14810 (30)
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 1 | 1
  Cycle 4 Day 1 |  |  | 32400 (NA) — There was 1 evaluable AUCtau measurement at this visit. | 42300 (NA) — There was 1 evaluable AUCtau measurement at this visit. |  | 17100 (NA) — There was 1 evaluable AUCtau measurement at this visit. | 58200 (NA) — There was 1 evaluable AUCtau measurement at this visit.

12. Secondary Outcome: Cycle 1 and Cycle 4 PF-07062119 PK Parameters: Area Under the Serum Concentration-Time Profile From Day 1 to Day 7 (168 Hours) (AUC168) - Priming Cohorts
Description: AUC168 was area under the serum concentration-time profile from Day 1 to Day 7 (168 hours) determined using linear/Log trapezoidal method.
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15 and Cycle 4 Day 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hour/mL
Arm/Group | Part 1A PF-07062119 400 µg/800 µg | Part 1A PF-07062119 400 µg/1200 µg | Part 1A PF-07062119 400 µg/1600 µg | Part 1A PF-07062119 400 µg/2100 µg | Part 1A PF-07062119 400 µg/2800 µg | PART 1A PF-07062119 400 µg/3700 µg | Part 1B PF-07062119 800 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + Bevacizumab 5 mg/kg Q2W-Priming
Number analyzed (Participants) | 10 | 6 | 6 | 8 | 4 | 4 | 4 | 4 | 3
ng•hour/mL
  Cycle 1 Day 1 | 2994 (51) | 2221 (57) | 3046 (53) | 4213 (61) | 4030 (26) | 4179 (31) | 3814 (33) | 4277 (48) | 3649 (20)
  Cycle 1 Day 15: number analyzed (Participants) | 9 | 6 | 6 | 8 | 4 | 4 | 4 | 3 | 3
  Cycle 1 Day 15 | 8971 (38) | 10570 (31) | 15660 (66) | 26700 (68) | 38220 (17) | 56500 (NA) — There was 1 evaluable AUC168 measurement at this visit. | 10950 (42) | 15540.785 (NA) — Two participants with evaluable AUC168 results at this visit (9980 and 24200 ng•hour/mL), so the geometric %CV was NA. | 18127.33 (NA) — Two participants with evaluable AUC168 results at this visit (15500 and 21200 ng•hour/mL), so the geometric %CV was NA.
  Cycle 4 Day 1: number analyzed (Participants) | 1 | 1 | 0 | 4 | 2 | 1 | 3 | 0 | 2
  Cycle 4 Day 1 | 22800 (NA) — There was 1 evaluable AUC168 measurement at this visit. | 31200 (NA) — There was 1 evaluable AUC168 measurement at this visit. |  | 95210 (17) | 117000 (NA) — Two participants with evaluable AUC168 results at this visit (117000 and 117000 ng•hour/mL), so the geometric %CV was NA. | 158000 (NA) — There was 1 evaluable AUC168 measurement at this visit. | 24754.80 (NA) — Two participants with evaluable AUC168 results at this visit (16000 and 38300 ng•hour/mL), so the geometric %CV was NA. |  | 50516.83 (NA) — Two participants with evaluable AUC168 results at this visit (47700 and 53500 ng•hour/mL), so the geometric %CV was NA.

13. Secondary Outcome: Cycle 1 and Cycle 4 PF-07062119 PK Parameters: AUC168 - Non-Priming Cohorts
Description: as for outcome 12
Time Frame: Cycle 1 Day 1 and Cycle 4 Day 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hour/mL
Arm/Group | Part 1A PF-07062119 45 µg | Part 1A PF-07062119 135 µg | Part 1A PF-07062119 400 µg | Part 1A PF-07062119 800 µg | Part 1A PF-07062119 1600 µg | Part 1B PF-07062119 400 µg Q2W + PF-06801591 300 mg Q4W | Part 1B PF-07062119 800 µg Q2W + Bevacizumab 5 mg/kg Q2W
Number analyzed (Participants) | 2 | 3 | 6 | 9 | 2 | 3 | 5
ng•hour/mL
  Cycle 1 Day 1 | 340.04 (NA) — Two participants with evaluable AUC168 results at this visit (298 and 388 ng•hour/mL), so the geometric %CV was NA. | 1209 (5) | 5564 (56) | 9041 (39) | 16500 (NA) — There was 1 evaluable AUC168 measurement at this visit. | 2684 (21) | 7133 (40)
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 1 | 1
  Cycle 4 Day 1 |  |  | 17400 (NA) — There was 1 evaluable AUC168 measurement at this visit. | 20700 (NA) — There was 1 evaluable AUC168 measurement at this visit. |  | 9830 (NA) — There was 1 evaluable AUC168 measurement at this visit. | 30900 (NA) — There was 1 evaluable AUC168 measurement at this visit.

14. Secondary Outcome: Pre-dose Trough Concentrations After Multiple Doses of PF-07062119
Description: PF-07062119 pre-dose trough concentrations were the serum PF-07062119 concentrations assessed at 0 min of Day 1 and Day 15 in each Cycle.
Time Frame: Cycle 1 Day 15, Cycle 2 Days 1 and 15, Cycle 3 Days 1 and 15, Cycle 4 Days 1 and 15, Cycle 5 Day 1, Cycle 8 Day 1 and Cycle 11 Day 1
Population: Analysis population included all enrolled participants who were treated and had at least 1 analyte concentration.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Part 1A PF-07062119 45 µg | Part 1A PF-07062119 135 µg | Part 1A PF-07062119 400 µg | Part 1A PF-07062119 800 µg | Part 1A PF-07062119 1600 µg | Part 1A PF-07062119 400 µg/800 µg | Part 1A PF-07062119 400 µg/1200 µg | Part 1A PF-07062119 400 µg/1600 µg | Part 1A PF-07062119 400 µg/2100 µg | Part 1A PF-07062119 400 µg/2800 µg | PART 1A PF-07062119 400 µg/3700 µg | Part 1B PF-07062119 400 µg Q2W + PF-06801591 300 mg Q4W | Part 1B PF-07062119 800 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 800 µg Q2W + Bevacizumab 5 mg/kg Q2W | Part 1B PF-07062119 1200 µg Q2W + Bevacizumab 5 mg/kg Q2W-Priming
Number analyzed (Participants) | 2 | 3 | 6 | 9 | 2 | 10 | 6 | 6 | 8 | 4 | 4 | 3 | 4 | 4 | 5 | 3
ng/mL
  Cycle 1 Day 15: number analyzed (Participants) | 2 | 3 | 5 | 8 | 0 | 9 | 6 | 6 | 8 | 4 | 4 | 3 | 4 | 3 | 5 | 3
  Cycle 1 Day 15 | 2.850 [2.77 to 2.93] | 8.140 [6.85 to 8.54] | 39.40 [31.7 to 48.1] | 56.95 [34.6 to 84.5] |  | 19.80 [12.9 to 42.0] | 22.55 [7.7 to 26.7] | 26.25 [19.5 to 36.0] | 25.30 [13.7 to 46.1] | 24.40 [19.8 to 29.4] | 30.40 [28.9 to 35.7] | 16.60 [14.7 to 19.5] | 29.80 [15.5 to 34.4] | 22.3 [20.0 to 25.5] | 44.20 [33.8 to 58.6] | 26.30 [21.2 to 26.6]
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 3 | 5 | 8 | 2 | 6 | 3 | 5 | 6 | 2 | 3 | 2 | 4 | 2 | 4 | 3
  Cycle 2 Day 1 | 3.265 [2.24 to 4.29] | 11.00 [10.8 to 12.1] | 68.50 [59.9 to 78.9] | 74.45 [30.3 to 113] | 47.40 [28.6 to 66.2] | 74.10 [48.3 to 84.4] | 69.80 [52.7 to 79.7] | 126.0 [65.4 to 226] | 176.5 [135 to 325] | 263.5 [230 to 297] | 242.0 [50.4 to 363] | 27.95 [25.3 to 30.6] | 57.70 [40.0 to 79.3] | 87.00 [86.6 to 87.4] | 63.25 [45.2 to 86.6] | 101.0 [92.1 to 109]
  Cycle 2 Day 15: number analyzed (Participants) | 1 | 1 | 4 | 6 | 1 | 4 | 1 | 3 | 5 | 2 | 1 | 2 | 4 | 2 | 4 | 3
  Cycle 2 Day 15 | 5.25 [5.25 to 5.25] | 14.5 [14.5 to 14.5] | 74.45 [71.7 to 79.0] | 91.45 [37.9 to 106] | 111.0 [111 to 111] | 94.40 [50.8 to 120] | 90.50 [90.5 to 90.5] | 100.0 [61.3 to 239] | 322.0 [221 to 427] | 432.0 [420 to 444] | 358.0 [358 to 358] | 35.6 [30.8 to 40.4] | 69.35 [26.1 to 129] | 54.80 [2.60 to 107] | 92.45 [81.0 to 125] | 153.0 [145 to 164]
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 1 | 1 | 3 | 1 | 1 | 1 | 2 | 4 | 2 | 1 | 1 | 3 | 0 | 3 | 2
  Cycle 3 Day 1 |  | 20.6 [20.6 to 20.6] | 80.2 [80.2 to 80.2] | 107.0 [101 to 110] | 129.0 [129 to 129] | 104.0 [104 to 104] | 110.0 [110 to 110] | 188.5 [0 to 377] | 414.0 [297 to 502] | 497.0 [489 to 505] | 528.0 [528 to 528] | 40.80 [40.8 to 40.8] | 72.10 [3.58 to 149] |  | 110.0 [63.0 to 132] | 181.5 [162 to 201]
  Cycle 3 Day 15: number analyzed (Participants) | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 4 | 2 | 1 | 1 | 3 | 0 | 2 | 2
  Cycle 3 Day 15 |  | 21.9 [21.9 to 21.9] | 82.1 [82.1 to 82.1] | 114.5 [105 to 124] | 76.90 [76.9 to 76.9] | 128.0 [128 to 128] | 130.0 [130 to 130] |  | 453.0 [312 to 517] | 542.5 [530 to 555] | 559.0 [559 to 559] | 36.40 [36.4 to 36.4] | 77.50 [0 to 189] |  | 150.5 [146 to 155] | 225.5 [204 to 247]
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 4 | 2 | 1 | 1 | 3 | 0 | 1 | 2
  Cycle 4 Day 1 |  |  | 74.9 [74.9 to 74.9] | 128.0 [113 to 143] | 133 [133 to 133] | 125.0 [125 to 125] | 162.0 [162 to 162] |  | 431.5 [377 to 541] | 528.5 [499 to 558] | 706.0 [706 to 706] | 37.20 [37.2 to 37.2] | 75.80 [0 to 205] |  | 141.0 [141 to 141] | 245.5 [216 to 275]
  Cycle 4 Day 15: number analyzed (Participants) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 2 | 2 | 1 | 1 | 3 | 0 | 1 | 1
  Cycle 4 Day 15 |  |  | 77.8 [77.8 to 77.8] | 122 [122 to 122] | 112 [112 to 112] | 108.0 [108 to 108] | 161.0 [161 to 161] |  | 429.5 [380 to 479] | 517.0 [512 to 522] | 795.0 [795 to 795] | 34.6 [34.6 to 34.6] | 94.40 [0 to 194] |  | 149.0 [149 to 149] | 226.0 [226 to 226]
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 1 | 2
  Cycle 5 Day 1 |  |  | 49.7 [49.7 to 49.7] | 117 [117 to 117] |  | 121.0 [121 to 121] |  |  | 357.0 [192 to 522] |  |  |  | 94.00 [0 to 180] |  | 147.0 [147 to 147] | 217.5 [189 to 246]
  Cycle 8 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Cycle 8 Day 1 |  |  |  |  |  |  |  |  | 517.5 [421 to 614] |  |  |  |  |  | 179.0 [179 to 179] | 125.0 [0 to 250]
  Cycle 11 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Cycle 11 Day 1 |  |  |  |  |  |  |  |  | 636.0 [636 to 636] |  |  |  |  |  | 189.0 [189 to 189] | 98.50 [0 to 197]

15. Secondary Outcome: Incidence of Anti-Drug Antibody (ADA) Positive Against PF-07062119
Description: Blood samples of approximately 4 mL, to provide a minimum of serum 2 mL, were collected for determination of ADA against PF-07062119. All samples were collected on Day 1 of a cycle (also on Day 15, in Cycle 1 only) and drawn pre-dose - within 6 hours prior to any of the drugs being administered. Starting at Cycle 5, blood samples for ADA against PF-07062119 were collected every 3rd cycle pre-dose (ie, Cycle 5 Day 1, Cycle 8 Day 1, Cycle 11 Day 1, etc.). Participants with an unresolved AE possibly related to ADA were asked to return to the clinic for ADA and drug concentration assessments at approximately 3 month intervals until the AE or its sequelae resolved or stabilized at a level acceptable to the investigator and sponsor up to a maximum of 9 months.
Time Frame: Pre-dose on Cycle 1 Day 1 and Day 15; Day 1 of Cycles 2 to 4; Day 1 of every 3rd cycle since Cycle 5
Population: Number of participants analyzed included all enrolled participants who received at least 1 dose of study intervention. Number analyzed refers to number of participants with ≥1 post-treatment ADA result.
Measure: Number; unit: Percentage
Arm/Group | Part 1A PF-07062119 45 µg | Part 1A PF-07062119 135 µg | Part 1A PF-07062119 400 µg | Part 1A PF-07062119 800 µg | Part 1A PF-07062119 1600 µg | Part 1A PF-07062119 400 µg/800 µg | Part 1A PF-07062119 400 µg/1200 µg | Part 1A PF-07062119 400 µg/1600 µg | Part 1A PF-07062119 400 µg/2100 µg | Part 1A PF-07062119 400 µg/2800 µg | PART 1A PF-07062119 400 µg/3700 µg | Part 1B PF-07062119 400 µg Q2W + PF-06801591 300 mg Q4W | Part 1B PF-07062119 800 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 800 µg Q2W + Bevacizumab 5 mg/kg Q2W | Part 1B PF-07062119 1200 µg Q2W + Bevacizumab 5 mg/kg Q2W-Priming
Number analyzed (Participants) | 2 | 3 | 6 | 9 | 2 | 10 | 6 | 6 | 8 | 4 | 4 | 3 | 4 | 4 | 5 | 3
Percentage
  Treatment-Induced: number analyzed (Participants) | 2 | 3 | 6 | 9 | 2 | 9 | 6 | 6 | 8 | 4 | 4 | 3 | 4 | 3 | 5 | 3
  Treatment-Induced | 0 | 0 | 16.7 | 11.1 | 0 | 0 | 0 | 16.7 | 0 | 25.0 | 25.0 | 0 | 25.0 | 33.3 | 20.0 | 66.7
  Treatment-Boosted: number analyzed (Participants) | 2 | 3 | 6 | 9 | 2 | 9 | 6 | 6 | 8 | 4 | 4 | 3 | 4 | 3 | 5 | 3
  Treatment-Boosted | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 25.0 | 0 | 0 | 0

16. Secondary Outcome: Titers of ADA Against PF-07062119
Description: Blood samples of approximately 4 mL, to provide a minimum of serum 2 mL, were collected for determination of ADA against PF-07062119. ADA titers of participants with positive PF-07062119 ADA (titer ≥70) are summarized.
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1 and End of Treatment
Population: Number of participants analyzed included all participants who had ≥1 post-treatment ADA result. Number analyzed refers to number of participants with ADA-positive samples (titer ≥70).
Measure: Median (Full Range); unit: titers
Arm/Group | Part 1A PF-07062119 45 µg | Part 1A PF-07062119 135 µg | Part 1A PF-07062119 400 µg | Part 1A PF-07062119 800 µg | Part 1A PF-07062119 1600 µg | Part 1A PF-07062119 400 µg/800 µg | Part 1A PF-07062119 400 µg/1200 µg | Part 1A PF-07062119 400 µg/1600 µg | Part 1A PF-07062119 400 µg/2100 µg | Part 1A PF-07062119 400 µg/2800 µg | PART 1A PF-07062119 400 µg/3700 µg | Part 1B PF-07062119 400 µg Q2W + PF-06801591 300 mg Q4W | Part 1B PF-07062119 800 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 800 µg Q2W + Bevacizumab 5 mg/kg Q2W | Part 1B PF-07062119 1200 µg Q2W + Bevacizumab 5 mg/kg Q2W-Priming
Number analyzed (Participants) | 2 | 3 | 6 | 9 | 2 | 9 | 6 | 6 | 8 | 4 | 4 | 3 | 4 | 3 | 5 | 3
titers
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Cycle 1 Day 1 |  |  |  |  |  |  |  |  |  | 326 [326 to 326] |  |  | 121 [121 to 121] |  |  |
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Cycle 1 Day 15 |  |  |  |  |  |  |  |  |  | 257 [257 to 257] |  |  | 540 [540 to 540] |  |  |
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Cycle 2 Day 1 |  |  |  | 197 [197 to 197] |  |  |  |  |  |  | 544 [544 to 544] |  | 427 [427 to 427] |  |  |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Cycle 3 Day 1 |  |  |  |  |  |  |  | 34295 [34295 to 34295] |  |  |  |  | 1063 [1063 to 1063] |  |  |
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Cycle 4 Day 1 |  |  |  |  |  |  |  | 439158 [439158 to 439158] |  |  |  |  | 16761 [16761 to 16761] |  |  |
  Cycle 5 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 5 Day 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 70 [70 to 70]
  Cycle 5 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 8 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 8 Day 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 140562 [140562 to 140562]
  Cycle 11 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Cycle 11 Day 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 120976 [206 to 241746]
  Cycle 14 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 14 Day 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 351572 [351572 to 351572]
  Cycle 17 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 17 Day 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 155181 [155181 to 155181]
  End of Treatment: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1
  End of Treatment |  |  | 4291 [4291 to 4291] |  |  |  |  |  |  | 392 [392 to 392] | 134678 [134678 to 134678] |  |  | 2413 [2413 to 2413] | 197 [197 to 197] | 344 [344 to 344]

17. Secondary Outcome: Incidence of Neutralizing Antibody (NAb) Positive Against PF-07062119
Description: Blood samples of approximately 4 mL, to provide a minimum of serum 2 mL, were collected for determination of NAb against PF-07062119. All samples were collected on Day 1 of a cycle (also on Day 15, in Cycle 1 only) and will be drawn pre-dose - within 6 hours prior to any of the drugs being administered. Starting at Cycle 5, blood samples for NAb against PF-07062119 were collected every 3rd cycle pre-dose (ie, Cycle 5 Day 1, Cycle 8 Day 1, Cycle 11 Day 1, etc). An NAb sample was defined as positive when NAb titer was ≥2.
Time Frame: Pre-dose on Cycle 1 Day 1 and Day 15; Day 1 of Cycles 2 to 4; Day 1 of every 3rd cycle since Cycle 5
Population: Number of participants analyzed included all enrolled participants who received at least 1 dose of study intervention. Number analyzed refers to number of participants with ≥1 post-treatment NAb result.
Measure: Number; unit: Percentage
Arm/Group | Part 1A PF-07062119 45 µg | Part 1A PF-07062119 135 µg | Part 1A PF-07062119 400 µg | Part 1A PF-07062119 800 µg | Part 1A PF-07062119 1600 µg | Part 1A PF-07062119 400 µg/800 µg | Part 1A PF-07062119 400 µg/1200 µg | Part 1A PF-07062119 400 µg/1600 µg | Part 1A PF-07062119 400 µg/2100 µg | Part 1A PF-07062119 400 µg/2800 µg | PART 1A PF-07062119 400 µg/3700 µg | Part 1B PF-07062119 400 µg Q2W + PF-06801591 300 mg Q4W | Part 1B PF-07062119 800 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 800 µg Q2W + Bevacizumab 5 mg/kg Q2W | Part 1B PF-07062119 1200 µg Q2W + Bevacizumab 5 mg/kg Q2W-Priming
Number analyzed (Participants) | 2 | 3 | 6 | 9 | 2 | 10 | 6 | 6 | 8 | 4 | 4 | 3 | 4 | 4 | 5 | 3
Percentage
  Treatment-Induced: number analyzed (Participants) | 2 | 3 | 6 | 9 | 2 | 9 | 6 | 6 | 8 | 4 | 4 | 3 | 4 | 3 | 5 | 3
  Treatment-Induced | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 16.7 | 0 | 25.0 | 25.0 | 0 | 25.0 | 33.3 | 0 | 66.7
  Treatment-Boosted: number analyzed (Participants) | 2 | 3 | 6 | 9 | 2 | 9 | 6 | 6 | 8 | 4 | 4 | 3 | 4 | 3 | 5 | 3
  Treatment-Boosted | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Incidence of ADA Positive Against PF-06801591
Description: Blood samples of approximately 4 mL, to provide a minimum of serum 2 mL, were collected for determination of ADA against PF-06801591. All samples were collected on Day 1 of a cycle (also on Day 15, in Cycle 1 only) and drawn pre-dose - within 6 hours prior to any of the drugs being administered. Starting at Cycle 5, blood samples for ADA against PF-06801591 in Part 1B were collected every 3rd cycle pre-dose (ie, Cycle 5 Day 1, Cycle 8 Day 1, Cycle 11 Day 1, etc). Participants with an unresolved AE possibly related to ADA were asked to return to the clinic for ADA and drug concentration assessments at approximately 3 month intervals until the AE or its sequelae resolved or stabilized at a level acceptable to the investigator and sponsor up to a maximum of 9 months. A participant was PF-06801591 ADA positive when ADA titer was ≥99.
Time Frame: Cycle 1 Day 1 and Day 15, Cycle 2 Day 1 and Day 15, Cycle 3 Day 1 and Day 15, Cycle 4 Day 15, Cycle 5 Day 15 and End of Treatment
Population: Analysis population included all participants who had ≥1 post-treatment ADA result.
Measure: Number; unit: Percentage
Arm/Group | Part 1B PF-07062119 400 µg Q2W + PF-06801591 300 mg Q4W | Part 1B PF-07062119 800 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + PF-06801591 300 mg Q4W-Priming
Number analyzed (Participants) | 3 | 4 | 1
Percentage | 0 | 0 | 0

19. Secondary Outcome: Percent Change From Baseline in Immune Biomarkers (CD3+ and CD8+ Cells/mm2 CT+, PD-L1 Tumor Cell Membrane Staining and PD-L1 Positive Immune Cells Per Tumor Area) in Pre-treatment and On-Treatment Paired Tumor Biopsies
Description: Tumor biospecimens from archival and/de novo biopsies were used to analyze candidate nucleic acid and protein and cellular biomarkers for their ability to inform those participants who were most likely to benefit from treatment with the study interventions. De novo tumor biopsies obtained during therapy and upon disease progression could be used to help confirm pharmacodynamic effects of treatment and investigate potential acquired mechanisms of resistance (ie, presence of but not limited to regulatory T-cells or myeloid derived suppressor cells and other immune suppressive cells or proteins).
Time Frame: Baseline (Baseline was defined as the time closest to, but prior to, the start of study drug administration in the first cycle), Cycle 3 Day 1
Population: Number of participants analyzed included all enrolled participants with at least 1 of the biomarkers evaluated at pre and/or post dose. Number analyzed refers to number of participants with non-missing test.
Measure: Median (Full Range); unit: Percentage
Arm/Group | Part 1A PF-07062119 45 µg | Part 1A PF-07062119 135 µg | Part 1A PF-07062119 400 µg | Part 1A PF-07062119 800 µg | Part 1A PF-07062119 1600 µg | Part 1A PF-07062119 400 µg/800 µg | Part 1A PF-07062119 400 µg/1200 µg | Part 1A PF-07062119 400 µg/1600 µg | Part 1A PF-07062119 400 µg/2100 µg | Part 1A PF-07062119 400 µg/2800 µg | PART 1A PF-07062119 400 µg/3700 µg | Part 1B PF-07062119 400 µg Q2W + PF-06801591 300 mg Q4W | Part 1B PF-07062119 800 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 800 µg Q2W + Bevacizumab 5 mg/kg Q2W | Part 1B PF-07062119 1200 µg Q2W + Bevacizumab 5 mg/kg Q2W-Priming
Number analyzed (Participants) | 2 | 3 | 6 | 9 | 2 | 10 | 6 | 6 | 8 | 4 | 3 | 3 | 4 | 4 | 4 | 3
Percentage
  CD3+ Cells/mm2 CT+ (cells/mm2): number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0
  CD3+ Cells/mm2 CT+ (cells/mm2) |  |  |  | -34.1 [-34.1 to -34.1] |  |  |  |  |  | 456.0 [89.1 to 822.8] | 482.2 [482.2 to 482.2] |  |  |  | 39.6 [39.6 to 39.6] |
  CD8+ Cells/mm2 CT+ (cells/mm2): number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0
  CD8+ Cells/mm2 CT+ (cells/mm2) |  |  |  | -23.3 [-23.3 to -23.3] |  |  |  |  |  | 1848.0 [290.7 to 3405.3] | 1378.5 [1378.5 to 1378.5] |  |  |  | 28.4 [28.4 to 28.4] |
  PD-L1 Tumor Cell Membrane Staining (%): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  PD-L1 Tumor Cell Membrane Staining (%) |  |  |  |  |  |  |  |  |  | 0 [0 to 0] | -100.0 [-100.0 to -100.0] |  |  |  |  |
  PD-L1 Positive Immune Cells per Tumor Area (%): number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
  PD-L1 Positive Immune Cells per Tumor Area (%) |  |  |  | 1500.0 [1500.0 to 1500.0] |  |  |  |  |  | -20.0 [-20.0 to -20.0] | 700.0 [700.0 to 700.0] |  |  |  | -100.0 [-100.0 to -100.0] |

20. Secondary Outcome: Number of Participants With Confirmed Objective Response
Description: Tumor assessments included all known or suspected disease sites. Imaging included contrast enhanced chest, abdomen and pelvis CT or MRI scans; brain CT or MRI scan for participants with known or suspected brain metastases; bone scan and/or bone x rays for participants with known or suspected bone metastases. For participants with known CT contrast allergy, a non-contrast CT of the chest with contrast enhanced abdominal and pelvic MRI could be used. The same imaging technique used to characterize each identified and reported lesion at baseline was employed in the tumor assessments. Assessment of response used Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Objective Response was defined as complete response (CR) + partial response (PR).
Time Frame: Baseline up to maximum of 4 years
Population: Analysis population included all enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A PF-07062119 45 µg | Part 1A PF-07062119 135 µg | Part 1A PF-07062119 400 µg | Part 1A PF-07062119 800 µg | Part 1A PF-07062119 1600 µg | Part 1A PF-07062119 400 µg/800 µg | Part 1A PF-07062119 400 µg/1200 µg | Part 1A PF-07062119 400 µg/1600 µg | Part 1A PF-07062119 400 µg/2100 µg | Part 1A PF-07062119 400 µg/2800 µg | PART 1A PF-07062119 400 µg/3700 µg | Part 1B PF-07062119 400 µg Q2W + PF-06801591 300 mg Q4W | Part 1B PF-07062119 800 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 800 µg Q2W + Bevacizumab 5 mg/kg Q2W | Part 1B PF-07062119 1200 µg Q2W + Bevacizumab 5 mg/kg Q2W-Priming
Number analyzed (Participants) | 2 | 3 | 6 | 9 | 2 | 10 | 6 | 6 | 8 | 4 | 4 | 3 | 4 | 4 | 5 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: 4 Years
Description: Same event may appear as both an AE and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both serious and non-serious event during the study. Safety analysis set included all participants who took at least 1 dose of study intervention.
Groups:
- Total: Overall Population
Arm/Group | Part 1A PF-07062119 45 µg | Part 1A PF-07062119 135 µg | Part 1A PF-07062119 400 µg | Part 1A PF-07062119 800 µg | Part 1A PF-07062119 1600 µg | Part 1A PF-07062119 400 µg/800 µg | Part 1A PF-07062119 400 µg/1200 µg | Part 1A PF-07062119 400 µg/1600 µg | Part 1A PF-07062119 400 µg/2100 µg | Part 1A PF-07062119 400 µg/2800 µg | Part 1A PF-07062119 400 µg/3700 µg | Part 1B PF-07062119 400 µg Q2W + PF-06801591 300 mg Q4W | Part 1B PF-07062119 800 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 1200 µg Q2W + PF-06801591 300 mg Q4W-Priming | Part 1B PF-07062119 800 µg Q2W + Bevacizumab 5 mg/kg Q2W | Part 1B PF-07062119 1200 µg Q2W + Bevacizumab 5 mg/kg Q2W-Priming | Total
All-Cause Mortality (participants affected / at risk) | 2/2 | 1/3 | 5/6 | 8/9 | 1/2 | 6/10 | 3/6 | 3/6 | 1/8 | 1/4 | 4/4 | 2/3 | 2/4 | 2/4 | 2/5 | 1/3 | 44/79
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/3 | 2/6 | 3/9 | 1/2 | 4/10 | 4/6 | 2/6 | 4/8 | 1/4 | 2/4 | 0/3 | 0/4 | 3/4 | 2/5 | 1/3 | 30/79
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3 | 6/6 | 9/9 | 2/2 | 10/10 | 5/6 | 6/6 | 8/8 | 4/4 | 4/4 | 3/3 | 4/4 | 4/4 | 5/5 | 3/3 | 78/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A PF-07062119 45 µg (N=2) | Part 1A PF-07062119 135 µg (N=3) | Part 1A PF-07062119 400 µg (N=6) | Part 1A PF-07062119 800 µg (N=9) | Part 1A PF-07062119 1600 µg (N=2) | Part 1A PF-07062119 400 µg/800 µg (N=10) | Part 1A PF-07062119 400 µg/1200 µg (N=6) | Part 1A PF-07062119 400 µg/1600 µg (N=6) | Part 1A PF-07062119 400 µg/2100 µg (N=8) | Part 1A PF-07062119 400 µg/2800 µg (N=4) | Part 1A PF-07062119 400 µg/3700 µg (N=4) | Part 1B PF-07062119 400 µg Q2W + PF-06801591 300 mg Q4W (N=3) | Part 1B PF-07062119 800 µg Q2W + PF-06801591 300 mg Q4W-Priming (N=4) | Part 1B PF-07062119 1200 µg Q2W + PF-06801591 300 mg Q4W-Priming (N=4) | Part 1B PF-07062119 800 µg Q2W + Bevacizumab 5 mg/kg Q2W (N=5) | Part 1B PF-07062119 1200 µg Q2W + Bevacizumab 5 mg/kg Q2W-Priming (N=3) | Total (N=79)
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 6
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rectal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 7
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A PF-07062119 45 µg (N=2) | Part 1A PF-07062119 135 µg (N=3) | Part 1A PF-07062119 400 µg (N=6) | Part 1A PF-07062119 800 µg (N=9) | Part 1A PF-07062119 1600 µg (N=2) | Part 1A PF-07062119 400 µg/800 µg (N=10) | Part 1A PF-07062119 400 µg/1200 µg (N=6) | Part 1A PF-07062119 400 µg/1600 µg (N=6) | Part 1A PF-07062119 400 µg/2100 µg (N=8) | Part 1A PF-07062119 400 µg/2800 µg (N=4) | Part 1A PF-07062119 400 µg/3700 µg (N=4) | Part 1B PF-07062119 400 µg Q2W + PF-06801591 300 mg Q4W (N=3) | Part 1B PF-07062119 800 µg Q2W + PF-06801591 300 mg Q4W-Priming (N=4) | Part 1B PF-07062119 1200 µg Q2W + PF-06801591 300 mg Q4W-Priming (N=4) | Part 1B PF-07062119 800 µg Q2W + Bevacizumab 5 mg/kg Q2W (N=5) | Part 1B PF-07062119 1200 µg Q2W + Bevacizumab 5 mg/kg Q2W-Priming (N=3) | Total (N=79)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 6
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 12
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 3 | 1 | 2 | 3 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 17
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 4 | 8 | 2 | 6 | 2 | 6 | 7 | 4 | 4 | 3 | 3 | 2 | 3 | 3 | 57
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 3 | 5 | 2 | 2 | 3 | 1 | 6 | 1 | 2 | 0 | 3 | 1 | 3 | 2 | 34
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 6
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Rectal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Small intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 5
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 7 | 2 | 2 | 1 | 0 | 6 | 1 | 1 | 0 | 2 | 3 | 1 | 1 | 29
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Axillary pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Chills (General disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 3 | 11
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 4 | 3 | 1 | 4 | 3 | 4 | 2 | 0 | 0 | 1 | 2 | 2 | 0 | 3 | 30
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Injection site discolouration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Injection site dryness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Injection site erythema (General disorders) | 1 | 1 | 6 | 5 | 0 | 5 | 2 | 3 | 2 | 2 | 1 | 1 | 2 | 1 | 4 | 1 | 37
Injection site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Injection site pruritus (General disorders) | 0 | 1 | 4 | 3 | 0 | 4 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 2 | 0 | 20
Injection site rash (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Injection site reaction (General disorders) | 1 | 1 | 0 | 1 | 0 | 2 | 3 | 1 | 3 | 1 | 2 | 1 | 2 | 3 | 0 | 2 | 23
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 11
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 6
Pre-existing condition improved (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 1 | 2 | 0 | 2 | 0 | 0 | 3 | 0 | 1 | 1 | 2 | 0 | 0 | 2 | 16
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 4 | 6 | 2 | 2 | 2 | 2 | 3 | 2 | 2 | 1 | 2 | 0 | 3 | 1 | 32
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacillus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Herpes simplex reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Injection related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 4
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 9
Amylase increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 5
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 9
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 8
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 4
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 9
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 9
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 3 | 1 | 0 | 4 | 2 | 1 | 2 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 20
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 5 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 15
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 7
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 10
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 5
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 6
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 3 | 0 | 1 | 3 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 15
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 3 | 2 | 1 | 0 | 2 | 2 | 1 | 0 | 17
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 3 | 1 | 3 | 1 | 0 | 0 | 0 | 1 | 15
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 5
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated on 10 October 2023. Study termination was due to a strategic decision but not any safety concerns or requests from any regulatory authorities. This BR presents the study results of dose escalation phase (Part 1) collected by the study completion date (28-Nov-2023). Dose expansion phase (Part 2) of the study was not conducted due to the study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT04171141/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT04171141/SAP_001.pdf